CLINICAL TRIAL: NCT00002764
Title: METASTASECTOMY AND CHEMOTHERAPY FOR LUNG METASTASES FROM SOFT TISSUE SARCOMA: A RANDOMIZED PHASE III STUDY (AN INTERGROUP STUDY WITH THE SCANDINAVIAN SARCOMA GROUP)
Brief Title: Surgery With or Without Combination Chemotherapy in Treating Patients With Lung Metastases From Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Eastern Cooperative Oncology Group (Network); Scandinavian Sarcoma Group (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-62933; EORTC-62933; E-EORTC-62933; SSG-EORTC-62933; SWOG-EORTC-62933
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Endometrial Cancer; Kidney Cancer; Metastatic Cancer; Ovarian Cancer; Pheochromocytoma; Sarcoma
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; recurrent adult soft tissue sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; localized benign pheochromocytoma; regional pheochromocytoma; lung metastases; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma; ovarian sarcoma; clear cell sarcoma of the kidney; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Kidney Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Pheochromocytoma; Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Sarcoma, Endometrial Stromal | interventions — Filgrastim; Doxorubicin; Ifosfamide

INTERVENTIONS:
Biological: filgrastim
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether surgery plus combination chemotherapy is more effective than surgery alone in treating patients with lung metastases from soft tissue sarcoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery plus combination chemotherapy with that of surgery alone in treating patients who have soft tissue sarcoma that has spread to the lung.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare disease control, overall survival, and relapse-free survival in patients with lung metastases secondary to soft tissue sarcoma treated with high-dose doxorubicin and ifosfamide with or without filgrastim (G-CSF) before and after metastasectomy vs metastasectomy alone. II. Determine the safety and morbidity of this regimen in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to location of metastases (unilateral vs bilateral). Patients are randomized to 1 of 2 treatment arms. Arm I: Patients are assigned to regimen A or B. Regimen A: Patients receive high-dose doxorubicin IV and ifosfamide IV continuously on day 1 and filgrastim (G-CSF) subcutaneously on days 3-13. Regimen B: Patients receive chemotherapy as above without G-CSF. Treatment on both regimens continues every 3 weeks for 3 courses. Patients then undergo radical pulmonary metastasectomy via thoracotomy or sternotomy with wedge resection or lobectomy. Patients with responding disease after metastasectomy receive 2 additional courses on the regimen to which they were originally assigned. Arm II: Patients undergo radical pulmonary metastasectomy as in arm I. Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 340 patients (170 per treatment arm) will be accrued for this study within approximately 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven soft tissue sarcoma with pulmonary metastases for which radical metastasectomy is feasible Eligible subtypes: Malignant fibrous histiocytoma Liposarcoma Synovial sarcoma Malignant paraganglioma Fibrosarcoma Leiomyosarcoma Neurogenic sarcoma Unclassified sarcoma Angiosarcoma (including hemangiopericytoma) Miscellaneous sarcoma (including mixed mesodermal tumors of the uterus) Ineligible subtypes: Alveolar rhabdomyosarcoma Kaposi's sarcoma Rhabdomyosarcoma of any type Malignant mesothelioma Chondrosarcoma Neuroblastoma Dermatofibrosarcoma Osteosarcoma Epithelioid sarcoma Primitive neuroectodermal tumor Ewing's sarcoma No extrapulmonary disease Previously treated local recurrence allowed Patients with primarily metastatic disease must have undergone radical treatment of primary tumor according to local protocols Reevaluation of metastases required before randomization

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 120,000/mm3 Hepatic: Bilirubin no greater than 1.25 times normal Renal: Creatinine no greater than 1.6 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of cardiovascular disease Other: No other severe medical illness (including psychosis) No prior or concurrent other primary malignancy except adequately treated carcinoma in situ of the cervix or basal cell carcinoma

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease Prior neoadjuvant or adjuvant chemotherapy for primary soft tissue sarcoma allowed if cumulative dose of doxorubicin no greater than 200 mg/m2 At least 1 year since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 1996-04; Primary Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A.N. Van Geel, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center; Ronald H. Blum, MD, Study Chair — NYU Langone Health; Thor A. Alvegard, MD, PhD, Study Chair — Lund University Hospital; Laurence H. Baker, DO, FACOI, Study Chair — University of Michigan Rogel Cancer Center
Locations (1):
- Lund University Hospital, Lund, Sweden